CLINICAL TRIAL: NCT03258645
Title: Pradaxa Initiation Post-Stroke Study: SITS-Pradaxa 1. A Retrospective Analysis From the SITS-AF Registry on Treatment Initiation of Dabigatran Etexilate in Non-valvular Atrial Fibrillation Patients Hospitalized With Acute Ischemic Stroke
Brief Title: This Study Uses the SITS Registry to Find Out When Patients With a Heart Rhythm Disorder (Atrial Fibrillation) Start Treatment With Dabigatran After They Had a Stroke
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Collaborators: Karolinska University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 1160.235
Record Dates: First submitted 2017-07-18; First posted 2017-08-23 (Actual); Results first posted 2020-07-09 (Actual); Last update posted 2020-07-09 (Actual); Status verified 2020-07

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Dabigatran

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Acute ischemic stroke: Non-valvular atrial fibrillation patients hospitalized with an acute ischemic stroke
  Interventions: Drug: Dabigatran

INTERVENTIONS:
Drug: Dabigatran — Oral anticoagulant (NOAC) thrombin inhibitor
  Other Names: Pradaxa

SUMMARY:
This is an observational study in patients with non-valvular atrial fibrillation (NVAF) presenting to the hospital with a first acute ischemic stroke based on existing data recorded in the SITS International Registry (located in Sweden) by physicians in several European countries, such as Italy, United Kingdom, Czech Republic, Sweden, Germany, Poland, Spain, Finland, Portugal, Slovakia, Denmark, Estonia, Norway Belgium, Hungary, Slovenia, Croatia, Austria, Lithuania, France, Greece, Netherlands, Ireland, Ukraine and Iceland.

The aim of this study is to explore the current real world use of dabigatran for stroke prevention in NVAF patients in the post-stroke setting. Secondary data from eligible European patients registered in the SITS registry will be considered; countries of origin are not known a priori.

ELIGIBILITY:
Inclusion criteria:

* Patients with non-valvular Atrial Fibrillation (NVAF)
* Patients presenting with their first acute ischemic stroke
* ≥18 years of age

Exclusion criteria:

- Documentation that the patient was enrolled or is planned to be enrolled in an investigational clinical trial at the time of the onset of the index event and for the duration of the data collection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1000
Sampling Method: Non-Probability Sample
Enrollment: 1489 (Actual)
Dates: Start 2018-11-15 (Actual); Primary Completion 2019-06-17 (Actual); Study Completion 2019-06-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- SITS International (c/o Karolinska University Hospital), Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Escudero-Martinez I, Mazya M, Teutsch C, Lesko N, Gdovinova Z, Barbarini L, Fryze W, Karlinski M, Kobayashi A, Krastev G, Paiva Nunes A, Pasztoova K, Peeters A, Sobolewski P, Vilionskis A, Toni D, Ahmed N; SITS Investigators. Dabigatran initiation in patients with non-valvular AF and first acute ischaemic stroke: a retrospective observational study from the SITS registry. BMJ Open. 2020 May 19;10(5):e037234. doi: 10.1136/bmjopen-2020-037234. PMID 32434935
- See also: Related Info — https://trials.boehringer-ingelheim.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This retrospective study using existing data from the Safe Implementation of Treatments in Stroke (SITS) International Stroke Registry assessed the timing of dabigatran treatment initiation in patients with non-valvular atrial fibrillation after the first ever ischemic stroke (3 months of follow-up thereafter) to prevent secondary stroke.
Pre-assignment Details: In this non-interventional study based on existing data, no patients were screened.
Groups:
- Total: Patients with non-valvular atrial fibrillation (NVAF) who were initiating dabigatran after hospitalization for first ever ischaemic stroke (the index event) in order to prevent secondary stroke based on existing data from the Safe Implementation of Treatments in Stroke (SITS) International Stroke Registry. Their follow-up period was around 3 months after the index event.
Period: Overall Study
Arm/Group | Total
Started | 1489
Completed | 1489
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Patients with non-valvular atrial fibrillation (NVAF) who were initiating dabigatran after hospitalization for first ever ischaemic stroke (the index event) in order to prevent secondary stroke in existing data from the Safe Implementation of Treatments in Stroke (SITS) International Stroke Registry.
Arm/Group | Total
Number analyzed (Participants) | 1489
Age, Continuous [Mean (Standard Deviation); unit: Years] | 75 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 788
  Male | 701
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Non-Valvular Atrial Fibrillation (NVAF) According to the Timing of Dabigatran Initiation After the First Ever Ischaemic Stroke (the Index Event)
Description: To evaluate the timing of dabigatran treatment initiation in patients with non-valvular atrial fibrillation (NVAF) after hospitalization for first ever ischaemic stroke (the index event) in order to prevent secondary stroke.
Time Frame: Up to 3 months of follow-up after index event
Population: Patients with non-valvular atrial fibrillation who were initiating dabigatran after hospitalization for first ever ischaemic stroke to prevent secondary stroke in existing data from the Safe Implementation of Treatments in Stroke International Stroke Registry. Analysis was on patients with dabigatran treatment initiation timing information only.
Measure: Number; unit: Percentage of participants
Arm/Group | Total
Number analyzed (Participants) | 1240
Percentage of participants
  0 - 24 hours (h) | 5.9
  > 24 - 72 h | 15.3
  > 3 - 7 days (d) | 27.7
  > 7 - 14 d | 33.1
  > 14 - 28 d | 14.0
  > 28 d - 3 months | 4.0

2. Secondary Outcome: National Institute of Health Stroke Scale (NIHSS) at First Ever Ischaemic Stroke According to Dabigatran Initiation Time Period
Description: The National Institute of Health Stroke Scale (NIHSS) score on patients with non-valvular atrial fibrillation and dabigatran initiation timing information. The NIHSS is a scale of stroke severity with 15 items and a score range from 0 to 42. 0 = no stroke; 1-4 = minor stroke; 5-15 = moderate stroke; 15-20 = moderate/severe stroke; 21-42 = severe stroke. Results were reported according to their dabigatran initiation timing categories.
Time Frame: At first ever ischaemic stroke (index event) date, up to 1 day.
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Score on a scale
Groups:
- 0 - 24 Hours: Patients with non-valvular atrial fibrillation (NVAF) who were initiating dabigatran after hospitalization for first ever ischaemic stroke (the index event) in order to prevent secondary stroke in existing data from the Safe Implementation of Treatments in Stroke (SITS) International Stroke Registry. Their follow-up period was around 3 months after the index event.
  Only patients with dabigatran initiation time less than 24 hours following index event were included in this group.
- > 24 - 72 Hours: Patients with non-valvular atrial fibrillation (NVAF) who were initiating dabigatran after hospitalization for first ever ischaemic stroke (the index event) in order to prevent secondary stroke in existing data from the Safe Implementation of Treatments in Stroke (SITS) International Stroke Registry. Their follow-up period was around 3 months after the index event.
  Only patients with dabigatran initiation time greater than 24 hours up to 72 hours following index event were included in this group.
- > 3 - 7 Days: Patients with non-valvular atrial fibrillation (NVAF) who were initiating dabigatran after hospitalization for first ever ischaemic stroke (the index event) in order to prevent secondary stroke in existing data from the Safe Implementation of Treatments in Stroke (SITS) International Stroke Registry. Their follow-up period was around 3 months after the index event.
  Only patients with dabigatran initiation time greater than 3 days up to 7 days following index event were included in this group.
- > 7 - 14 Days: Patients with non-valvular atrial fibrillation (NVAF) who were initiating dabigatran after hospitalization for first ever ischaemic stroke (the index event) in order to prevent secondary stroke in existing data from the Safe Implementation of Treatments in Stroke (SITS) International Stroke Registry. Their follow-up period was around 3 months after the index event.
  Only patients with dabigatran initiation time greater than 7 days up to 14 days following index event were included in this group.
- > 14 - 28 Days: Patients with non-valvular atrial fibrillation (NVAF) who were initiating dabigatran after hospitalization for first ever ischaemic stroke (the index event) in order to prevent secondary stroke in existing data from the Safe Implementation of Treatments in Stroke (SITS) International Stroke Registry. Their follow-up period was around 3 months after the index event.
  Only patients with dabigatran initiation time greater than 14 days up to 28 days following index event were included in this group.
- > 28 Days - 3 Months: Patients with non-valvular atrial fibrillation (NVAF) who were initiating dabigatran after hospitalization for first ever ischaemic stroke (the index event) in order to prevent secondary stroke in existing data from the Safe Implementation of Treatments in Stroke (SITS) International Stroke Registry. Their follow-up period was around 3 months after the index event.
  Only patients with dabigatran initiation time greater than 28 days up to 3 months following index event were included in this group.
Arm/Group | 0 - 24 Hours | > 24 - 72 Hours | > 3 - 7 Days | > 7 - 14 Days | > 14 - 28 Days | > 28 Days - 3 Months
Number analyzed (Participants) | 73 | 190 | 344 | 410 | 174 | 49
Score on a scale | 8 [5 to 14] | 8 [5 to 14] | 8 [6 to 13] | 12 [7 to 17] | 14 [10 to 18] | 15 [9 to 19]
Statistical Analysis 1: Comparison: 0 - 24 Hours vs > 24 - 72 Hours vs > 3 - 7 Days vs > 7 - 14 Days vs > 14 - 28 Days vs > 28 Days - 3 Months; Univariate linear regression with the continuous dependent variable of time-to-initiation for dabigatran in days and independent variable of National Institute of Health Stroke Scale (NIHSS) score at index date was applied; Test type: Other; p < 0.001, Regression, Linear

3. Secondary Outcome: Previous Modified Rankin Scale (mRS) at First Ever Ischaemic Stroke According to Dabigatran Initiation Time Period
Description: Previous Modified Rankin Scale (mRS) collected at first ever ischaemic stroke (index event). The Modified Rankin scale (mRS) is Scored as follows: 0 = No symptoms, 1 = No significant disability. Able to carry out all usual activities, despite some symptoms, 2 = Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities, 3 = Moderate disability. Requires some help, but able to walk unassisted, 4 = Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted, 5 = Severe disability. Requires constant nursing care and attention, bedridden, incontinent, 6 = Death. Higher scores indicate worse outcome. Results were reported according to their dabigatran initiation timing categories.
Time Frame: At first ever ischaemic stroke (index event) date, up to 1 day.
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Score on a scale
Arm/Group | 0 - 24 Hours | > 24 - 72 Hours | > 3 - 7 Days | > 7 - 14 Days | > 14 - 28 Days | > 28 Days - 3 Months
Number analyzed (Participants) | 73 | 190 | 344 | 410 | 174 | 49
Score on a scale | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 1]
Statistical Analysis 1: Comparison: 0 - 24 Hours vs > 24 - 72 Hours vs > 3 - 7 Days vs > 7 - 14 Days vs > 14 - 28 Days vs > 28 Days - 3 Months; Univariate linear regression with the continuous dependent variable of time-to-initiation for dabigatran in days and independent variable of Modified Rankin Scale (mRS) at index date was applied; Test type: Other; p = 0.01, Regression, Linear

4. Secondary Outcome: Age of Patients According to Dabigatran Initiation Time Period
Description: Age of patients according to their start dabigatran time period. Results were reported according to their dabigatran initiation timing categories. CHA2DS2-VASc and HAS-BLED were used in the statistical analysis. CHA2DS2-VASc is the Congestive heart failure, Hypertension, Age (> 75), Diabetes mellitus, Stroke/transient ischemic attack(TIA), Vascular disease, Age 65-74, Sex Category score. HAS-BLED is the Hypertension, Abnormal renal and liver function, Stroke (1 point), Bleeding history or predisposition, Labile international normalised ratio (INR), Elderly (>65 years), Drugs and Alcohol Score.
Time Frame: At first ever ischaemic stroke (index event), up to 1 day.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Years
Arm/Group | 0 - 24 Hours | > 24 - 72 Hours | > 3 - 7 Days | > 7 - 14 Days | > 14 - 28 Days | > 28 Days - 3 Months
Number analyzed (Participants) | 73 | 190 | 344 | 410 | 174 | 49
Years | 72 (11) | 74 (10) | 75 (9) | 75 (9) | 76 (9) | 77 (10)
Statistical Analysis 1: Comparison: 0 - 24 Hours vs > 24 - 72 Hours vs > 3 - 7 Days vs > 7 - 14 Days vs > 14 - 28 Days vs > 28 Days - 3 Months; Multivariate linear regression with the continuous dependent variable of time-to-initiation for dabigatran in days and independent variable of age, Diastolic blood pressure (DBP), CHA2DS2-VASc, HAS-BLED, and History/Predisposition To Bleeding at index date was applied; Test type: Other — CHA2DS2-VASc is the Congestive heart failure, Hypertension, Age (> 75), Diabetes mellitus, Stroke/TIA, Vascular disease, Age 65-74, Sex Category score. HAS-BLED is the Hypertension, Abnormal renal and liver function, Stroke (1 point), Bleeding history or predisposition, Labile INR, Elderly (>65 years), Drugs and Alcohol Score; p = 0.016, Regression, Linear; Relation between age and dabigatran initiation time was reported; Odds Ratio (OR) = 1.13, 95% CI 2-sided [1.02 to 1.25]

5. Secondary Outcome: Diastolic Blood Pressure (DBP) of Patients According to Dabigatran Initiation Time Period
Description: Diastolic blood pressure (DBP) of patients according to their start dabigatran time period. Results were reported according to their dabigatran initiation timing categories.
Time Frame: At first ever ischaemic stroke (index event), up to 1 day.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: millimetre of mercury (mm Hg)
Arm/Group | 0 - 24 Hours | > 24 - 72 Hours | > 3 - 7 Days | > 7 - 14 Days | > 14 - 28 Days | > 28 Days - 3 Months
Number analyzed (Participants) | 73 | 190 | 344 | 410 | 174 | 49
millimetre of mercury (mm Hg) | 87 (12) | 83 (15) | 84 (14) | 85 (15) | 85 (17) | 91 (16)
Statistical Analysis 1: Comparison: 0 - 24 Hours vs > 24 - 72 Hours vs > 3 - 7 Days vs > 7 - 14 Days vs > 14 - 28 Days vs > 28 Days - 3 Months; [analysis description as in outcome 4, analysis 1]; Test type: Other — [test comment as in outcome 4, analysis 1]; p = 0.002, Regression, Linear; Relation between Diastolic blood pressure (DBP) and dabigatran initiation time was reported; Odds Ratio (OR) = 1.12, 95% CI 2-sided [1.04 to 1.21]

6. Secondary Outcome: CHA2DS2-VASc of Patients According to Dabigatran Initiation Time Period
Description: The Congestive heart failure, Hypertension, Age (> 75), Diabetes mellitus, Stroke/TIA, Vascular disease, Age 65-74, Sex Category (CHA2DS2-VASc) score of patients according to their start dabigatran time period. CHA2DS2-VASc is used to determine the need for an anticoagulation therapy, relating the high scores to a great risk of stroke and a low score corresponds to a lower risk of stroke. CHA2DS2-VASc stroke risk score ranges from 0 to 9 with 0 being the best outcome. Results were reported according to their dabigatran initiation timing categories.
Time Frame: At first ever ischaemic stroke (index event), up to 1 day.
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Score on a scale
Arm/Group | 0 - 24 Hours | > 24 - 72 Hours | > 3 - 7 Days | > 7 - 14 Days | > 14 - 28 Days | > 28 Days - 3 Months
Number analyzed (Participants) | 73 | 190 | 344 | 410 | 174 | 49
Score on a scale | 5 [4 to 6] | 5 [4 to 6] | 5 [4 to 6] | 5 [4 to 6] | 5 [4 to 6] | 5 [4 to 6]
Statistical Analysis 1: Comparison: 0 - 24 Hours vs > 24 - 72 Hours vs > 3 - 7 Days vs > 7 - 14 Days vs > 14 - 28 Days vs > 28 Days - 3 Months; [analysis description as in outcome 4, analysis 1]; Test type: Other — [test comment as in outcome 4, analysis 1]; p = 0.04, Regression, Linear; Relation between CHA2DS2-VASc and dabigatran initiation time was reported; Odds Ratio (OR) = 1.10, 95% CI 2-sided [1.00 to 1.21]

7. Secondary Outcome: HAS-BLED of Patients According to Dabigatran Initiation Time Period
Description: The Hypertension, Abnormal renal and liver function, Stroke (1 point), Bleeding history or predisposition, Labile INR, Elderly (>65 years), Drugs and Alcohol (HAS-BLED) Score of patients according to their start dabigatran time period. HAS-BLED score ranges from 0 to 9 with higher scores indicating greater risk of bleeding. Results were reported according to their dabigatran initiation timing categories.
Time Frame: At first ever ischaemic stroke (index event), up to 1 day.
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Score on a scale
Arm/Group | 0 - 24 Hours | > 24 - 72 Hours | > 3 - 7 Days | > 7 - 14 Days | > 14 - 28 Days | > 28 Days - 3 Months
Number analyzed (Participants) | 73 | 190 | 344 | 410 | 174 | 49
Score on a scale | 3 [2 to 3] | 3 [2 to 3] | 3 [2 to 3] | 3 [2 to 3] | 3 [2 to 3] | 3 [2 to 3]
Statistical Analysis 1: Comparison: 0 - 24 Hours vs > 24 - 72 Hours vs > 3 - 7 Days vs > 7 - 14 Days vs > 14 - 28 Days vs > 28 Days - 3 Months; [analysis description as in outcome 4, analysis 1]; Test type: Other — [test comment as in outcome 4, analysis 1]; p = 0.051, Regression, Linear; Relation between HAS-BLED and dabigatran initiation time was reported; Odds Ratio (OR) = 0.90, 95% CI 2-sided [0.45 to 1.00]

8. Secondary Outcome: Percentage of Patients With History of or Predisposition to Bleeding According to Dabigatran Initiation Time Period
Description: Percentage of patients with History of or predisposition to bleeding according to their start dabigatran time period. Results were reported according to their dabigatran initiation timing categories.
Time Frame: At first ever ischaemic stroke (index event), up to 1 day.
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | 0 - 24 Hours | > 24 - 72 Hours | > 3 - 7 Days | > 7 - 14 Days | > 14 - 28 Days | > 28 Days - 3 Months
Number analyzed (Participants) | 73 | 190 | 344 | 410 | 174 | 49
Percentage of participants | 2.1 | 1.1 | 3.0 | 3.0 | 1.8 | 4.4
Statistical Analysis 1: Comparison: 0 - 24 Hours vs > 24 - 72 Hours vs > 3 - 7 Days vs > 7 - 14 Days vs > 14 - 28 Days vs > 28 Days - 3 Months; [analysis description as in outcome 4, analysis 1]; Test type: Other — [test comment as in outcome 4, analysis 1]; p = 0.026, Regression, Linear; Relation between History/Predisposition To Bleeding and dabigatran initiation time was reported; Odds Ratio (OR) = 0.91, 95% CI 2-sided [0.9 to 0.93]

9. Secondary Outcome: Number of Times of Reason to Delay Oral Anticoagulation (OAC) Entered by Physicians.
Description: Number of time the corresponding reason to delay oral anticoagulation (OAC) entered by physicians. More than one reasons could be entered for each patient. Index event was defined as the first ever acute ischemic stroke that led to hospital admission for eligible patients.
Time Frame: Up to 3 months of follow-up after index event.
Population: Patients with non-valvular atrial fibrillation who were initiating dabigatran after first ever ischaemic stroke to prevent secondary stroke in existing data from the Safe Implementation of Treatments in Stroke International Stroke Registry. Analysis was on patients with dabigatran initiation timing information and non-missing endpoint results.
Measure: Number; unit: Times
Arm/Group | Total
Number analyzed (Participants) | 203
Times
  Haemorrhagic transformation | 40
  Intracranial Haemorrhage (ICH) Spontaneous | 8
  Severity Infarct | 61
  Size of Infarct | 52
  Location Infarct | 14
  Intervention used to treat ischemic stroke | 8
  Altered coagulation parameters | 5
  Patients bleeding risk factors | 18
  Patients stroke risk factors | 6
  Patient preference | 4
  Recommendation from specialist | 6
  Practical considerations | 14
  Reason is not specified | 27
  Other reasons | 5

10. Secondary Outcome: Number of Times of Reason to Delay Dabigatran Initiation Entered by Physicians According to Dabigatran Initiation Time Period
Description: Physicians' reason to delay dabigatran initiation according to their start dabigatran time period. More than one reasons could be entered for each patient. Index event was defined as the first ever acute ischemic stroke that led to hospital admission for eligible patients.
Time Frame: At first ever ischaemic stroke (index event), up to 1 day.
Population: as for outcome 9
Measure: Number; unit: Times
Arm/Group | 0 - 24 Hours | > 24 - 72 Hours | > 3 - 7 Days | > 7 - 14 Days | > 14 - 28 Days | > 28 Days - 3 Months
Number analyzed (Participants) | 1 | 2 | 6 | 26 | 42 | 10
Times
  Haemorrhagic transformation | 0 | 0 | 2 | 2 | 8 | 1
  Intracranial Haemorrhage (ICH) pontaneous | 0 | 0 | 0 | 1 | 3 | 0
  Severity Infarct | 0 | 0 | 1 | 7 | 12 | 2
  Size of Infarct | 0 | 0 | 2 | 9 | 12 | 3
  Location Infarct | 0 | 0 | 0 | 3 | 2 | 0
  Intervention used to treat ischemic stroke | 0 | 0 | 0 | 2 | 3 | 0
  Altered coagulation parameters | 0 | 0 | 0 | 2 | 1 | 0
  Patients bleeding risk factors | 0 | 1 | 0 | 4 | 6 | 0
  Patients stroke risk factors | 0 | 0 | 0 | 2 | 2 | 1
  Recommendation from specialist | 0 | 0 | 0 | 0 | 2 | 1
  Practical considerations | 1 | 1 | 0 | 0 | 3 | 3
  Reason is not specified | 0 | 0 | 1 | 5 | 4 | 1
  Other reasons | 0 | 0 | 0 | 0 | 1 | 0

11. Secondary Outcome: Number of Times of Reason to Chose Daily Dosage of 220 Milligram of Dabigatran Entered by Physicians
Description: Number of times of corresponding reason of choosing daily dosage of 220 milligram of dabigatran entered by physicians. More than one reasons could be entered for each patient. Index event was defined as the first ever acute ischemic stroke that led to hospital admission for eligible patients.
Time Frame: Up to 3 months of follow-up after index event.
Population: as for outcome 9
Measure: Number; unit: Times
Arm/Group | Total
Number analyzed (Participants) | 382
Times
  Haemorrhagic transformation | 6
  Intracranial Haemorrhage (ICH) spontaneous | 3
  Severity of stroke | 18
  Size of infarct | 13
  Location of infarct | 8
  Intervention used to treat stroke | 4
  Altered coagulation parameters | 7
  Patients bleeding risk | 6.3
  Patients stroke risk | 27
  Recommendation from specialist | 32
  Reason is not specified | 95
  Other reasons | 10
  Patients age | 209
  Co-medication | 11
  Co-morbidities | 16
  Renal function | 48

12. Secondary Outcome: Number of Times of Reason to Chose Daily Dosage of 300 Milligram of Dabigatran Entered by Physicians
Description: Number of times the corresponding reason for choosing daily dosage of 300 milligram of dabigatran entered by physicians. More than one reasons could be entered for each patient. Index event was defined as the first ever acute ischemic stroke that led to hospital admission for eligible patients.
Time Frame: Up to 3 months of follow-up after index event.
Population: as for outcome 9
Measure: Number; unit: Times
Arm/Group | Total
Number analyzed (Participants) | 475
Times
  Intracranial Haemorrhage (ICH) spontaneous | 1
  Severity of stroke | 38
  Size of infarct | 16
  Location of infarct | 18
  Intervention used to treat stroke | 3
  Altered coagulation parameters | 10
  Patients bleeding risk | 34
  Patients stroke risk | 89
  Recommendation from specialist | 50
  Reason is not specified | 216
  Other reasons | 1
  Patients age | 139
  Co-medication | 5
  Co-morbidities | 19
  Renal function | 47

ADVERSE EVENTS:
Time Frame: Adverse event information was not applicable for this study.
Description: As this is a observational study with existing data from the Safe Implementation of Treatments in Stroke (SITS) International Stroke Registry, safety monitoring and safety reporting on an individual case level is not applicable.
Arm/Group | Total
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
This is an observational study on existing data. All findings are conditional on a selected sample of subjects who had initiated treatment prior to dying, having a second stroke or leaving care.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results.

Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days.

BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2017-07-05): https://cdn.clinicaltrials.gov/large-docs/45/NCT03258645/Prot_000.pdf
  • Statistical Analysis Plan (2018-11-07): https://cdn.clinicaltrials.gov/large-docs/45/NCT03258645/SAP_001.pdf